CLINICAL TRIAL: NCT04209088
Title: Interest of Pulmonary Ultrasound to Predict Evolution Towards Bronchopulmonary Dysplasia in Premature Infants at Gestational Age Less Than or Equal to 34 Weeks of Gestation
Acronym: PREDYSPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 87RI19_0023 (PREDYSPE)
Record Dates: First submitted 2019-12-20; First posted 2019-12-23 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: bronchopulmonary dysplasia; premature newborn; ultrasonography
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulmonary ultrasounds (Experimental): All patients will be included in the experimental arm
  Interventions: Other: Pulmonary ultrasounds

INTERVENTIONS:
Other: Pulmonary ultrasounds — Two ultrasounds will be performed by the same pediatrician for each child included: the first at nine days of life +/- two days, the second at fifteen days of life +/- two days.
  A blind replay of ultrasound images to calculate the score will be performed by a another investigator.

SUMMARY:
Each year, between 50,000 and 60,000 children are born prematurely in France. Among them, 10% are born at 26 - 30 week's gestation and 5% are born before 26 week's gestation.

Bronchopulmonary dysplasia (BPD) affects at least one-quarter of infants born with a birth weight less than 1500 grams.

BPD is defined by the need for oxygen after 28 days of life in any children born prematurely. In addition, the severity of BPD can be categorized as mild (room air tolerated at 36 weeks), moderate (oxygen requirement between 22 and 29 %) and severe (oxygen requirement 30% or need for ventilation support).

Bronchopulmonary dysplasia is responsible for significant respiratory morbidity and impaired neurological outcomes.

Pulmonary imaging such as tomodensitometry, MRI or scintigraphy can be abnormal and therefore coud theorically be helpful for an early diagnosis. Unfortunatelly, theses examinations are irradiating, expensive or difficult to perform in an everyday practice. Therefore lung imaging for BPD diagnosis. Is not recommanded in current official guidelines.

Pulmonary ultrasound has already been studied in premature newborns. A pilot study carried out on 21 patients showed that pulmonary ultrasonography at one and two weeks of life could predict the risk of bronchopulmonary dysplasia. The score used in this study was the LUS score previously validated by Brat et al. Advantages of this examination are to be non-invasive and easily performed at the patient's bedside. Nevertheless this study focused on a small population with a low number of moderate / severe dysplasia.

In addition, Czernik et al. have highlighted that the index of myocardial performance of the right ventricle was increased at seven and ten days of life in children who subsequently developed BPD.

The investigators propose in this study to evaluate a new prediction score for DBP, the modified LUS score, associating the LUS score with an echographic evaluation of the right heart (myocardial performance index).

ELIGIBILITY:
Inclusion Criteria:

* Premature neonates with gestational age less than or equal to 34 weeks of amenorrhea.
* Hospitalized in the NICU or neanatology unit at Limoges University Hospital at day 9 +/- 2 and day 15 +/- 2 of life
* participation agreement of at least one of the parents.

Exclusion Criteria:

* Cardiac malformations
* Congenital lung malformation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2020-05-29 (Actual); Primary Completion 2023-06-06 (Estimated); Study Completion 2023-06-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate the AUC of the modified LUS score to predict the occurrence of BPD | Day 9

SECONDARY OUTCOMES:
Evaluate the AUC of the modified LUS score to predict the occurrence of BPD | Day 15
Concordance of measured LUS scores between operator and reviewer | Day 9
Concordance of measured LUS scores between operator and reviewer | Day 15

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Limoges, France

IPD SHARING:
Plan to Share IPD: No